CLINICAL TRIAL: NCT06958445
Title: The Efficacy of Sodium Alginate on Prevention of Oral Mucositis and Quality of Life for Patients With Breast Cancer Undergoing Adjuvant Radiotherapy
Brief Title: Prevention of Oral Mucositis and Improvement of Quality of Life for Patients With Breast Cancer Undergoing Adjuvant Radiotherapy
Acronym: SAFE
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Yi-Sheng Chou, Physician, Taipei City Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TCHIRB-11211009
Record Dates: First submitted 2025-04-24; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Breast Carcinoma
Keywords: breast cancer; adjuvant radiotherapy; esophagitis; mucositis; alginate
MeSH Terms: conditions — Breast Neoplasms; Esophagitis; Mucositis | interventions — Alginates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esophagitis prevention (Experimental): Patients are taking orally alginos suspension 10cc qid on Monday to Friday during the course of radiotherapy
  Interventions: Drug: Alginos Oral Suspension
- Control (No Intervention): Patients are not taking any medications during the course of radiotherapy

INTERVENTIONS:
Drug: Alginos Oral Suspension — containing: Sodium alginate 50mg/mL Sodium bicarbonate 26.7mg/mL Calcium carbonate 16mg/mL
  Other Names: alginate; sodium alginate
  Arms: Esophagitis prevention

SUMMARY:
Breast cancer patients receiving adjuvant radiotherapy after surgery, particularly when the supraclavicular lymph nodes are included in the treatment area, frequently experience side effects of esophagitis such as sore throat, hoarseness, difficulty swallowing, and a reduction in white blood cell counts. Currently, no specific treatments exist to mitigate these adverse effects. This study proposes the use of alginate as a potential solution to alleviate these symptoms and improve the quality of life in breast cancer patients undergoing radiotherapy.

Although the side effects of radiotherapy do not typically pose a clinical risk, they have a profound impact on patients' quality of life, particularly affecting nutrition intake and well-being. This study aims to evaluate whether alginate can prevent these radiotherapy-induced side effects and improve the overall quality of life for breast cancer patients.

The trial will be conducted with 150 breast cancer patients undergoing adjuvant radiotherapy after surgery. The patients will receive 10cc of alginate orally, four times daily. Weekly evaluations will be conducted to assess the presence and improvement of symptoms such as sore throat, hoarseness, difficulty swallowing, and changes in white blood cell counts. Quality of life will be measured using the EORTC BR23 and QLQ-C30 questionnaires at the first and last sessions of radiation therapy.

The study aims to determine whether alginate can effectively prevent the side effects of radiation therapy, such as oral inflammation, sore throat, hoarseness, difficulty swallowing, and a decrease in blood cell counts. Furthermore, it will evaluate whether these improvements lead to a better quality of life for breast cancer patients undergoing adjuvant radiotherapy.

DETAILED DESCRIPTION:
Breast cancer patients receiving adjuvant radiotherapy after surgery, particularly when the supraclavicular lymph nodes are included in the treatment area, frequently experience side effects of esophagitis such as sore throat, hoarseness, difficulty swallowing, and a reduction in white blood cell counts. Currently, no specific treatments exist to mitigate these adverse effects. This study proposes the use of alginate as a potential solution to alleviate these symptoms and improve the quality of life in breast cancer patients undergoing radiotherapy.

While the use of alginate for preventing radiation-induced esophagitis is under-explored, two existing studies suggest promising outcomes. The first study, conducted in Japan in 1990. However, a second study involving 39 patients demonstrated that administering alginate (10-15cc) four times daily during radiation therapy reduced the severity of oral inflammation. Although the side effects of radiotherapy do not typically pose a clinical risk, they have a profound impact on patients' quality of life, particularly affecting nutrition intake and well-being. This study aims to evaluate whether alginate can prevent these radiotherapy-induced side effects and improve the overall quality of life for breast cancer patients.

1. Study Design: The trial will be conducted with 150 breast cancer patients undergoing adjuvant radiotherapy after surgery. The patients will receive 10cc of alginate orally, four times daily. Weekly evaluations will be conducted to assess the presence and improvement of symptoms such as sore throat, hoarseness, difficulty swallowing, and changes in white blood cell counts. Quality of life will be measured using the EORTC BR23 and QLQ-C30 questionnaires at the first and last sessions of radiation therapy.
2. Inclusion and Exclusion Criteria I.Inclusion Criteria: Patients over 18 years of age. Diagnosed with breast cancer with metastatic lymphadenopathy undergoing adjuvant radiotherapy.Willing to participate in the alginate treatment trial.

   II.Exclusion Criteria: Concurrent chemotherapy during radiation therapy. Cognitive impairment or inability to respond to questionnaire content.Requirement for a low-sodium diet.Conditions such as heart failure, renal insufficiency
3. Recruitment and Consent Process:

   Eligible patients will be invited to participate during their routine clinic visits. The principal investigator will explain the study protocol in detail, ensuring the patients fully understand the trial. Upon providing signed informed consent, the patients will be enrolled in the study.
4. Clinical Endpoints:

   I.Primary Endpoint: Evaluation of changes in the quality of life using the EORTC BR23 and QLQ-C30 questionnaires.

   II.Secondary Endpoint: The assessment of radiation therapy side effects, including oral inflammation, sore throat, hoarseness, difficulty swallowing, and a decrease in blood cell counts, as measured by the Common Terminology Criteria for Adverse Events (CTCAE) scale.

   III.Tertiary Endpoints: Evaluation of miRNA and cytokine profile in patient's serum
5. Expected Outcomes The study aims to determine whether alginate can effectively prevent the side effects of radiation therapy, such as oral inflammation, sore throat, hoarseness, difficulty swallowing, and a decrease in blood cell counts. Furthermore, it will evaluate whether these improvements lead to a better quality of life for breast cancer patients undergoing adjuvant radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Diagnosed with female breast cancer with metastatic lymphadenopathy undergoing adjuvant radiotherapy.
* Willing to participate in the alginate treatment trial.

Exclusion Criteria:

* Concurrent chemotherapy during radiation therapy.
* Cognitive impairment or inability to respond to questionnaire content.
* Requirement for a low-sodium diet.
* Conditions such as heart failure, renal insufficiency

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who have breast cancer
Enrollment: 90 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of Quality of Life Using a Validated Questionnaire | "From enrollment to the end of treatment at 7 weeks
  The validated questionnaire incorporates the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 and its associated quality of life (QoL) module designed to assess QoL during adjuvant radiotherapy. "QLQ" refers to the Quality of Life Questionnaire. The breast cancer-specific module, QLQ-BR23, is used in conjunction with the core QLQ-C30 instrument. Together, the QLQ-C30 and QLQ-BR23 comprise a total of 53 questions. The instruments include five multi-item scales designed to evaluate body image, sexual functioning, systemic therapy side effects, breast symptoms, and arm symptoms. These items are rated on a 4-point Likert scale (1 = "not at all" to 4 = "very much"). Additionally, single items assess sexual enjoyment, future perspective, and distress caused by hair loss. Higher scores on these symptom scales indicate greater symptom burden. In contrast, questions 29 and 30 assess overall health and overall quality of life, respectively.

SECONDARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | From enrollment to the end of treatment at 7 weeks
  Side effects including oral inflammation, sore throat, hoarseness, difficulty swallowing, anemia, leukopenia, neutropenia, thrombocytopenia, mucositis and esophgitis

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Sheng Chou, M.D, Principal Investigator — Taipei City Hospital
Locations (1):
- Taipei City Hospital, Renai Branch, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] West K, Schneider M, Wright C, Beldham-Collins R, Coburn N, Tiver K, Gebski V, Stuart KE. Radiation-induced oesophagitis in breast cancer: Factors influencing onset and severity for patients receiving supraclavicular nodal irradiation. J Med Imaging Radiat Oncol. 2020 Feb;64(1):113-119. doi: 10.1111/1754-9485.12943. Epub 2019 Sep 4. PMID 31486274
- [Background] Upadhyay R, Bazan JG. Advances in Radiotherapy for Breast Cancer. Surg Oncol Clin N Am. 2023 Jul;32(3):515-536. doi: 10.1016/j.soc.2023.03.002. PMID 37182990
- [Background] Weber WP, Hanson SE, Wong DE, Heidinger M, Montagna G, Cafferty FH, Kirby AM, Coles CE. Personalizing Locoregional Therapy in Patients With Breast Cancer in 2024: Tailoring Axillary Surgery, Escalating Lymphatic Surgery, and Implementing Evidence-Based Hypofractionated Radiotherapy. Am Soc Clin Oncol Educ Book. 2024 Jun;44(3):e438776. doi: 10.1200/EDBK_438776. PMID 38815195
- [Background] Yu H, Lam KO, Green MD, Wu H, Yang L, Wang W, Jin J, Hu C, Wang Y, Jolly S, Spring Kong FM. Significance of radiation esophagitis: Conditional survival assessment in patients with non-small cell lung cancer. J Natl Cancer Cent. 2021 Feb 18;1(2):31-38. doi: 10.1016/j.jncc.2021.02.003. eCollection 2021 Jun. PMID 39035770
- [Background] Saldi S, Perrucci E, Fulcheri CPL, Mariucci C, Chierchini S, Ingrosso G, Falcinelli L, Podlesko AM, Merluzzi M, Bini V, Aristei C. Zinc-L-carnosine prevented dysphagia in breast cancer patients undergoing adjuvant radiotherapy: Results of a phase III randomized trial. Breast J. 2020 Sep;26(9):1882-1884. doi: 10.1111/tbj.13855. Epub 2020 May 7. No abstract available. PMID 32383225
- [Background] Fiets WE, van Helvoirt RP, Nortier JW, van der Tweel I, Struikmans H. Acute toxicity of concurrent adjuvant radiotherapy and chemotherapy (CMF or AC) in breast cancer patients. a prospective, comparative, non-randomised study. Eur J Cancer. 2003 May;39(8):1081-8. doi: 10.1016/s0959-8049(03)00178-3. PMID 12736107
- [Background] Gay HA, Oh JH, Apte AP, Daly MD, Adkins DR, Rich J, Oppelt PJ, Dyk PT, Mullen DF, Eschen L, Chin RI, Nussenbaum B, Haughey BH, Thorstad WL, Deasy JO. Predictors of acute throat or esophageal patient reported pain during radiation therapy for head and neck cancer. Clin Transl Radiat Oncol. 2018 Sep 4;13:1-6. doi: 10.1016/j.ctro.2018.08.004. eCollection 2018 Nov. PMID 30211324